CLINICAL TRIAL: NCT00332332
Title: Canadian Assessment of Patient Outcomes and Effectiveness of Enbrel (Etanercept) in Psoriasis
Brief Title: Canadian Assessment of Patient Outcomes and Effectiveness of Etanercept (Enbrel) in Psoriasis
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Amgen (Industry)
Collaborators: Wyeth is now a wholly owned subsidiary of Pfizer (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 20050180
Record Dates: First submitted 2006-05-30; First posted 2006-06-01 (Estimated); Results first posted 2011-06-14 (Estimated); Last update posted 2014-07-25 (Estimated); Status verified 2014-07

CONDITIONS: Psoriasis
Keywords: Phase IV; Psoriasis; Inflammation
MeSH Terms: conditions — Psoriasis; Inflammation | interventions — Etanercept

ARMS (1):
- etanercept (Experimental): Open label etanercept 50 mg twice weekly subcutaneously (SC) for 3 months followed by 50 mg twice a week week SC for 9 months, for a total treatment period of 12 months.
  Interventions: Biological: etanercept

INTERVENTIONS:
Biological: etanercept — etanercept subcutaneous injection
  Other Names: ENBREL

SUMMARY:
The purpose of this study is to evaluate the use of etanercept (Enbrel®) in the treatment of psoriasis in patients for a period of up to 1 year.

ELIGIBILITY:
Inclusion Criteria:

* 18 years of age or older at baseline
* Moderate to severe plaque psoriasis at baseline with a rating of moderate, marked or severe on the Physician Global Assessment (score of 3, 4 or 5)
* Able to start Enbrel (Etanercept) therapy per the approved product monograph

Exclusion Criteria

* Active infections at the initiation of Enbrel therapy.
* Evidence of skin conditions (i.e. eczema) other than psoriasis that would interfere with evaluations of the effect of study medication on psoriasis.
* Psoralen plus ultraviolet A radiation (PUVA) within 4 weeks or ultraviolet light B (UVB) therapy within 2 weeks of study drug initiation.
* Oral retinoids, cyclosporine, methotrexate, or any other systemic anti-psoriasis therapy within 4 weeks or efalizumab (Raptiva®) within 8 weeks of study drug initiation and during the study period.
* Topical Vitamin A or D analog preparations, or anthralin within 2 weeks of study drug initiation and during the study period.
* Have received Remicade® (infliximab), Humira® (adalimumab) or Amevive®(alefacept) within 3 months before the initiation of study medication or during the study period.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 246 (Actual)
Dates: Start 2006-03; Primary Completion 2009-07 (Actual); Study Completion 2010-02 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: MD, Study Director — Amgen

REFERENCES:
- [Background] Vender R, Lynde C, Gilbert M, Ho V, Sapra S, Poulin-Costello M. One-year, multicenter, open-label, single-arm study evaluating the safety and effectiveness of etanercept for the treatment of moderate-to-severe plaque psoriasis in a Canadian population. J Cutan Med Surg. 2013 Mar-Apr;17(2):129-38. doi: 10.2310/7750.2012.12036. PMID 23582167
- [Background] Vender R, Lynde C, Gilbert M, Ho V, Sapra S, Poulin-Costello M. Etanercept improves quality of life outcomes and treatment satisfaction in patients with moderate to severe plaque psoriasis in clinical practice. J Cutan Med Surg. 2012 Nov-Dec;16(6):407-16. doi: 10.1177/120347541201600609. PMID 23149196
- See also: AmgenTrials clinical trials website — http://www.amgentrials.com

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Participants were enrolled from 17 March 2006 through 30 June 2008
Groups:
- Etanercept: Open label etanercept administered subcutaneously at 50 mg twice weekly for 3 months, followed by a maintenance dose of 50 mg once weekly for the remaining 9 months of the study.
Period: Overall Study
Arm/Group | Etanercept
Started | 246
Received Study Medication | 230
Completed | 178
Not Completed | 68
Not completed — Adverse Event | 13
Not completed — Death | 1
Not completed — Withdrawal by Subject | 8
Not completed — Physician Decision | 1
Not completed — Lost to Follow-up | 3
Not completed — Protocol deviation | 4
Not completed — Noncompliance | 2
Not completed — Disease progression | 2
Not completed — Other | 18
Not completed — Did not receive study treatment | 16

BASELINE CHARACTERISTICS:
Arm/Group | Etanercept
Number analyzed (Participants) | 230
Age, Continuous [Mean (Standard Deviation); unit: Years] | 45.5 (11.5)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 95
  Male | 135
Race/Ethnicity, Customized [Number; unit: Participants]
  Caucasian | 215
  Black | 1
  Asian | 10
  American Indian or Alaska Native | 1
  Aborigine | 1
  Other | 2
Patient Global Assessment [Mean (Standard Deviation); unit: Units on a scale] — Patient global assessment of psoriasis scores range from 0 (good) to 5 (severe)
  Units on a scale | 4.0 (0.8)
Body Surface Area [Mean (Standard Deviation); unit: m^2] — Body surface area affected by psoriasis
  m^2 | 27.4 (21.3)
Dermatology Quality of Life Index Total Score [Mean (Standard Deviation); unit: Units on a scale] — This score ranges from 0 to 30, with 0 = no effect and 30 = large effect
  Units on a scale | 13.7 (6.1)

OUTCOME MEASURES:

1. Primary Outcome: Participants With a Status of Mild or Better on Physician Global Assessment at Month 12
Description: The number of participants with a status of mild or better (score of 0, 1 or 2) on the Physician Global Assessment (PGA) of psoriasis at Month 12. This scale ranges from 0 to 5, with 0 = best outcome.
Time Frame: Month 12
Population: Full Analysis Set, composed of enrolled participants who received at least one dose of study medication and who had a baseline and at least one post-baseline measurement of the endpoint of interest. Missing post-baseline values were imputed using last observation carried forward.
Measure: Number; unit: Participants
Arm/Group | Etanercept
Number analyzed (Participants) | 226
Participants | 166
Statistical Analysis 1: Comparison: Etanercept; Test type: Superiority or Other; Percentage of participants = 73.5, 95% CI [67.2 to 79.1]

2. Secondary Outcome: Percent Change From Baseline to Month 12 in Patient Global Assessment
Description: Percent change from Baseline to Month 12 in the Patient Global Assessment of psoriasis score. This score ranged from 0 (good) to 5 (severe). A negative change from Baseline indicates improvement in disease activity.
Time Frame: Baseline and Month 12
Population: Full Analysis Set, composed of enrolled participants who received at least one dose of study medication and who had a baseline and at least one post-baseline measurement of the endpoint of interest, with imputation using Last Observation Carried Forward (LOCF).
Measure: Mean (95% Confidence Interval); unit: Percent change
Arm/Group | Etanercept
Number analyzed (Participants) | 223
Percent change | -57.9 [-62.6 to -53.2]

3. Secondary Outcome: Percent Change From Baseline to Month 12 in Body Surface Area Affected by Psoriasis
Description: Percent change from Baseline to Month 12 in body surface area (BSA) affected by psoriasis. A reduction (indicated by a negative percent change from Baseline) in the BSA affected is indicative of improvement in disease activity.
Time Frame: Baseline and Month 12
Population: as for outcome 2
Measure: Mean (95% Confidence Interval); unit: Percent change
Arm/Group | Etanercept
Number analyzed (Participants) | 226
Percent change | -69.9 [-75.1 to -64.6]

4. Secondary Outcome: Percent Change From Baseline to Month 12 in the Dermatology Life Quality Index Total Score
Description: Percent change from Baseline to Month 12 in the Dermatology Life Quality Index (DLQI) total score. This score ranges from 0 to 30, where 0 = no effect and 30 = large effect. A reduction in DLQI total score is indicative of improvement in quality of life as it relates to the participant's psoriasis, and a negative change from Baseline indicates improvement.
Time Frame: Baseline and Month 12
Population: as for outcome 2
Measure: Mean (95% Confidence Interval); unit: Percent change
Arm/Group | Etanercept
Number analyzed (Participants) | 225
Percent change | -68.2 [-73.7 to -62.8]

ADVERSE EVENTS:
Time Frame: Up to 13 months
Description: The table of Other Adverse Events summarizes the most frequent non-serious occurrences of adverse events.
Arm/Group | Etanercept
Serious Adverse Events (participants affected / at risk) | 12/230
Other Adverse Events (participants affected / at risk) | 59/230
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Etanercept (N=230)
Atrial flutter (Cardiac disorders) | 1
Cardiac failure congestive (Cardiac disorders) | 1
Intestinal obstruction (Gastrointestinal disorders) | 1
Death (General disorders) | 1
Cellulitis (Infections and infestations) | 1
Sepsis (Infections and infestations) | 1
Subdural haematoma (Injury, poisoning and procedural complications) | 1
Diabetes mellitus inadequate control (Metabolism and nutrition disorders) | 1
Fluid retention (Metabolism and nutrition disorders) | 1
Basal cell carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1
Squamous cell carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1
Thyroid adenoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1
Thyroid gland cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1
Convulsion (Nervous system disorders) | 1
Pulmonary oedema (Respiratory, thoracic and mediastinal disorders) | 1
Erythema multiforme (Skin and subcutaneous tissue disorders) | 1
Aortic stenosis (Vascular disorders) | 1
Hypertension (Vascular disorders) | 1
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Etanercept (N=230)
Nasopharyngitis (Infections and infestations) | 18
Upper respiratory tract infection (Infections and infestations) | 16
Headache (Nervous system disorders) | 16
Psoriasis (Skin and subcutaneous tissue disorders) | 13

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
The Clinical Trial Agreement generally does not restrict an investigator's discussion of trial results after completion. The Agreement permits Amgen a limited period of time to review material discussing trial results (typically up to 45 days and possible extension). Amgen may remove confidential information, but authors have final control and approval of publication content. For multicenter studies, the investigator agrees not to publish any results before the first multi-center publication.